CLINICAL TRIAL: NCT03204097
Title: 1% Alendronate and Aloevera Gel Local Host Modulating Agents in Chronic Periodontitis Subjects With Class II Furcation Defects: A Randomized Controlled Clinical Trial
Brief Title: Local Host Modulating Agents Alendronate & Aloe Vera for Treatment of Furcation Defects in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and HOD, Dept of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2015-2016IP
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- group 1 (Placebo Comparator): Scaling and root planing (SRP) followed by placebo gel local drug delivery
  Interventions: Drug: placebo
- group 2 (Active Comparator): SRP followed by 1% Alendronate (ALN) gel
  Interventions: Drug: Alendronate
- group 3 (Active Comparator): SRP followed by Aloevera (AV) gel
  Interventions: Drug: Aloe Vera

INTERVENTIONS:
Drug: placebo — Oral prophylaxis followed by placement of placebo gel
  Other Names: inactive drug
  Arms: group 1
Drug: Alendronate — Oral prophylaxis followed by placement of Alendronate gel
  Other Names: ALN
  Arms: group 2
Drug: Aloe Vera — Oral prophylaxis followed by placement of Aloe Vera gel
  Other Names: AV
  Arms: group 3

SUMMARY:
Alendronate (ALN), commonly use bisphosphonates is proposed to have osteostimulative properties in vivo and in vitro, as shown by an increase in the matrix formation, and acts as a potent inhibitor of bone resorption. AV widely known for its wound healing, analgesic, antioxidant, antibacterial, antiviral, antifungal, immune boosting and significant anti-inflammatory properties. The present study aims to explore the efficacy of 1% ALN and AV gel as a local drug delivery as an adjunct to scaling and root planing (SRP) for the treatment of degree II furcation defects

DETAILED DESCRIPTION:
Alendronate (ALN), commonly use bisphosphonates is proposed to have osteostimulative properties in vivo and in vitro, as shown by an increase in the matrix formation, and acts as a potent inhibitor of bone resorption. AV widely known for its wound healing, analgesic, antioxidant, antibacterial, antiviral, antifungal, immune boosting and significant anti-inflammatory properties. The present study aims to explore the efficacy of 1% ALN and AV gel as a local drug delivery as an adjunct to scaling and root planing (SRP) for the treatment of degree II furcation defects.

Methods: Ninety patients with mandibular buccal class II furcation defects were randomly allocated into three treatment groups: SRP plus placebo gel (group 1), SRP plus 1% ALN gel (group 2) and SRP plus AV gel (group3). Clinical and radiographic parameters were recorded at baseline and gel were delivered at respective site. Then again all clinical and radiographic parameters were recorded after 6 and 12 months from baseline.

ELIGIBILITY:
Inclusion Criteria:Systemically healthy patients with mandibular class II furcation defects and asymptomatic endodontically vital mandibular molars with radiolucency in furcation area with PD ≥ 5mm and horizontal PD ≥ 3mm and with no history of antibiotic or any periodontal therapy in past 6 months were included in the study -

Exclusion Criteria:Subjects with any known systemic disease, allergic to alendronate or aloe vera, on systemic alendronate therapy, alcoholics, tobacco users, pregnant or lactating women

-

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in Bone defect depth | baseline, 6 & 12 months
  Assessed in percentage

SECONDARY OUTCOMES:
Change in modified sulcus bleeding index | baseline, 6 & 12 months
  scale 0-3
Change in Plaque index | baseline, 6 & 12 months
  scale 0-3
Change in pocket probing depth | baseline, 6 & 12 months
  measured in mm
Change in relative vertical clinical attachment level | baseline, 6 & 12 months
  measured in mm
Change in relative horizontal clinical attachment level | baseline, 6 & 12 months
  measured in mm